CLINICAL TRIAL: NCT03823495
Title: Effectiveness of a Peer-led Pain Management Program in Relieving Chronic Pain and Enhancing Pain Self-efficacy Among Older Adults: a Clustered Randomized Controlled Trial
Brief Title: Effectiveness of a Peer-led Pain Management Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PLPMP
Record Dates: First submitted 2018-09-12; First posted 2019-01-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Randomized Controlled Trial
Keywords: pain management; nursing home; elderly; non-drug
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 12-week PAP (one 1-hour session per week). Each session includes 20-minute exercise, 30-minute interactive pain management education, practices on non-drug management techniques, and portfolio entry for activities of the day.
  Interventions: Other: 12-week PAP
- Control group (No Intervention): The control group will receive the usual care and a pain management pamphlet distributed by nursing home staff

INTERVENTIONS:
Other: 12-week PAP — It is a non-drug intervention, using exercises to reduce elderlies chronic pain.
  Arms: Experimental group

SUMMARY:
Objective: To evaluate the efficacy of a peer-led pain management program (PAP) in improving pain self-efficacy, reduce pain, enhancing use of drugs and non-drug methods and quality of life among nursing home residents

Hypothesis: PAP lead by peer volunteer (PV) is more effective than receive usual care and pain management pamphlet, in reducing pain intensity, enhancing pain self-efficacy, use of drugs and non-drug methods, health-related quality of life upon completion of the PAP (week 12) and over time (week 24).

Design and subjects: Clustered randomized controlled trial with nursing homes as cluster; 288 residents will be recruited from 12 nursing homes. Each nursing home will be randomly allocated to experimental group (PV led PAP), control group (receive usual care and pain management pamphlet).

Study instruments: Brief Pain Inventory, Pain Self-Efficacy Questionnaire, Use of drugs and non-drug methods log book, Short Form Health Survey-12 and process evaluation.

Intervention: 12-week PAP (one 1-hour session per week).

Outcome measures: Pain intensity, pain self-efficacy, use of non-drug pain relief methods, perceived health-related quality of life and experience in participating PAP, to be collected at baseline (T0), week 12 (T1), and week 24 (T2).

Data analysis: Multilevel regression and/or Generalized Estimating Equation will be used for within-group and between- group comparisons.

Expected results: Significant reduction in pain and enhancement in pain-related parameters, making peers support models in elderly care.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of a peer-led pain management program (PAP) in improving pain self-efficacy, reduce pain, enhancing use of drugs and non-drug methods and quality of life among nursing home residents

Hypothesis: PAP lead by peer volunteer (PV) is more effective than receive usual care and pain management pamphlet, in reducing pain intensity, enhancing pain self-efficacy, use of drugs and non-drug methods, health-related quality of life upon completion of the PAP (week 12) and over time (week 24).

Design and subjects: Clustered randomized controlled trial with nursing homes as cluster; 288 residents will be recruited from 12 nursing homes. Each nursing home will be randomly allocated to experimental group (PV led PAP), control group (receive usual care and pain management pamphlet).

Study instruments: Brief Pain Inventory, Pain Self-Efficacy Questionnaire, Use of drugs and non-drug methods log book, Short Form Health Survey-12 and process evaluation.

Intervention: 12-week PAP (one 1-hour session per week). Each session includes 20-minute exercise, 30-minute interactive pain management education, practices on non-drug management techniques, and portfolio entry for activities of the day. The interventionist is the PV. The one hour session per week will consisted of 20-minute exercise, include correct body posture and alignment, stretching of arms, legs, and body muscles, balancing exercise; shoulder & neck exercise; knee exercise; towel dancing. While the 30-minute interactive pain management education as well as practices on non-drug management techniques. Topics include: 1) pain situations among older adults; effects of pain in daily life; can we do something? 2) The use of oral drugs for pain: effects and side-effects; 3) The use of non-drug therapy: hot pad & cold pad; how to use & safety issues? 4) The use of non-drug therapy: listening to music; 5) the use of non-drug therapy: massage; 6) the use of non-drug therapy: visual stimulation - watching the natural environment & making a photo album; 7) the use of non-drug therapy: sense of smell & taste- making a bag of dried flowers & tasting tea; 8) Revision & wrapping up. Portfolio entry include the PV will work with the participants to make entry on the activity of the day in the portfolio.

Outcome measures: Pain intensity, pain self-efficacy, use of non-drug pain relief methods, perceived health-related quality of life and experience in participating PAP, to be collected at baseline (T0), week 12 (T1), and week 24 (T2).

Data analysis: Multilevel regression and/or Generalized Estimating Equation will be used for within-group and between- group comparisons.

Expected results: Significant reduction in pain and enhancement in pain-related parameters, making peers support models in elderly care.

ELIGIBILITY:
Inclusion Criteria:

* scored ≥ 6 in the Abbreviated Mental Test Chinese Version
* scored ≥ 4 in the Brief Pain Inventory Chinese Version
* scored ≥ 60 in the Modified Barthel Index Chinese Version
* able to speak and understand Cantonese

Exclusion Criteria:

* scored ≥ 8 in the Geriatric Depression Scale Chinese Version
* history of psychotic disorders
* currently undergoing cancer treatment
* has conditions that limit safe participation in exercising

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2018-06-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Intensity (questionnaire) | Change from baseline to 12-week (after the intervention) and 24-week (follow up)
  Brief Pain Inventory is a 10 point likert scale ranging from 0 to 10. It will be used to assess the multidimensional nature of the participants' pain, including its intensity and subsequent interference with life activities

SECONDARY OUTCOMES:
Pain self-efficacy questionnaire (questionnaire) | Change from baseline to 12-week (after the intervention) and 24-week (follow up)
  Pain self-efficacy questionnaire is a 7-point likert scale ranging from 0 to 6. It will be used to assess the participants' confidence in their ability to perform specific tasks or their confidence in performing more generalized constructs such as coping with chronic non-malignant pain.
Use of drugs and non-drug methods | Change from baseline to 12-week (after the intervention) and 24-week (follow up)
  The drugs that are used, and their frequency of use will be collected from medication charts
Perceived health-related quality of life | Change from baseline to 12-week (after the intervention) and 24-week (follow up)
  The chinese version of the SF-12 questionnaire is a likert scale to assess participants perceived physical and mental health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tse MMY, Tang SK, Ng S, Li Y, Cheung DSK, Kwan RYC. Assessing the fidelity of a peer-led chronic pain management program (PAP). Trials. 2021 Sep 20;22(1):644. doi: 10.1186/s13063-021-05599-6. PMID 34544469
- [Derived] Tse MMY, Ng SSM, Lee PH, Bai X, Lo R, Tang SK, Chan KL, Li Y. Effectiveness of a Peer-Led Pain Management Program in Relieving Chronic Pain and Enhancing Pain Self-Efficacy Among Older Adults: A Clustered Randomized Controlled Trial. Front Med (Lausanne). 2021 Aug 5;8:709141. doi: 10.3389/fmed.2021.709141. eCollection 2021. PMID 34422864